CLINICAL TRIAL: NCT06268483
Title: Effect of Hyaluronic Acid Oral Supplementation on Sexual and Urinary Symptoms of Women With Recurrent Urinary Tract Infections
Acronym: JalUrol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JalUrol; Policlinico (Other: IRCCS Fondazione Ca' Granda Ospedale Maggiore Policlinico)
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Urinary Tract Infections, Recurrent
Keywords: urinary tract infection; hyaluronic acid
MeSH Terms: conditions — Urinary Tract Infections | interventions — Acetylglucosamine; Ascorbic Acid; Mannose; Propolis; Curcumin; Frankincense

STUDY DESIGN:
Intervention Model Description: randomized, crossover
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral supplementation of hyaluronic acid + anti-inflammatory (Active Comparator): Group I: an oral preparation (capsule) of HA 100 mg, CS 400 mg, N-Acetylglucosamine 200 mg and vitamin C 80 mg once a day in the morning plus an oral preparation of cranberry, D-mannose, propolis extract, tumeric and Boswellia twice a day for three months
  Interventions: Dietary Supplement: HA 100 mg, CS 400 mg, N-Acetylglucosamine 200 mg and vitamin C 80 mg + cranberry, D-mannose, propolis extract, tumeric and Boswellia; Dietary Supplement: cranberry, D-mannose, propolis extract, tumeric and Boswellia
- Anti-inflammatori (Active Comparator): Group C: an oral preparation of cranberry, D-mannose, propolis extract, tumeric and Boswellia twice a day for three months.
  Interventions: Dietary Supplement: HA 100 mg, CS 400 mg, N-Acetylglucosamine 200 mg and vitamin C 80 mg + cranberry, D-mannose, propolis extract, tumeric and Boswellia; Dietary Supplement: cranberry, D-mannose, propolis extract, tumeric and Boswellia

INTERVENTIONS:
Dietary Supplement: HA 100 mg, CS 400 mg, N-Acetylglucosamine 200 mg and vitamin C 80 mg + cranberry, D-mannose, propolis extract, tumeric and Boswellia — Group I: an oral preparation (capsule) of HA 100 mg, CS 400 mg, N-Acetylglucosamine 200 mg and vitamin C 80 mg once a day in the morning plus an oral preparation of cranberry, D-mannose, propolis extract, tumeric and Boswellia twice a day for three months.
Dietary Supplement: cranberry, D-mannose, propolis extract, tumeric and Boswellia — Group C: an oral preparation of cranberry, D-mannose, propolis extract, tumeric and Boswellia twice a day for three months.

SUMMARY:
Uncomplicated urinary tract infections (UTI) are one of the most common bacterial infections globally, causing a significant proportion of medical consultations in primary and outpatient settings. Recurrent UTI (rUTI) have a detrimental impact on the patient's quality of life, causing a negative effect on women's social relationships, self-esteem, as well as irritability and tiredness. Moreover, several real-life studies have shown that reproductive-aged women with rUTI more frequently experience sexual dysfunction as compared to controls without infections. The glycosaminoglycan layer of the bladder urothelium, mainly composed by chondroitin sulfate (CS) and hyaluronic acid (HA), provides a protective barrier against the penetration of bacteria. A deficiency of this layer facilitates bacterial adherence, leading to recurrent infection. Treatment to restore this layer with intravesical instillation of HA has been proven to reduce the incidence of rUTI episodes. Furthermore, intravesical instillation with HA has been associates with sexual function improvement in women with rUTI and painful bladder . Therefore, in conditions where the glycosaminoglycan layer of the bladder is impaired, such as rUTIs, treatment with HA to restore it appears to have a beneficial effect on urinary and sexual symptoms.

Recently, a randomized control trial has demonstrated that an oral formulation of HA, CS, quercetin and curcumin was effective in improving urinary symptoms in women undergoing intravesical chemotherapy for bladder cancer. However, there are no studies investigating the impact of the oral administration of HA and CS on the sexual and urinary symptoms of women with rUTI. Since rUTI are highly prevalent in sexually active women and exert a detrimental impact on women's quality of life, sexual and urinary symptoms, the identification of oral treatments that could alleviate these bothersome consequences is of primary clinical importance.

Therefore we will conduct this randomized, cross-over trial to evaluate the efficacy of an oral preparation of HA, CS, N-Acetylglucosamine and vitamin C in improving sexual and urinary symptoms in a cohort of reproductive-aged women with rUTI.

Methods:

Pre-menopausal, sexually active women referred to our center for symptomatic rUTIs. At the time of enrollment, participants were randomized with a 1:1 allocation ratio by means of a computer-generated random list in two groups: intervention (I) and control (C) (Figure 1).

Inclusion and exclusion criteria We included sexually active, reproductive-aged women with symptomatic rUTIs. Exclusion criteria: younger than 18, if they had used combined hormonal contraception during the previous 6 months; pregnant, breastfeeding or trying to conceive, if they had symptoms of upper UTI, a history of urinary tract anomalies/vesicoureteral reflux, stress urinary incontinence, interstitial cystitis, diabetes, urinary tract stones, neurologic conditions, clinical depression or depressive symptoms.

All women will be assessed with a thorough medical and sexual history. To psychometrically quantify sexual function impairment all participants completed The Female Sexual Function Index (FSFI) questionnaire at baseline and at each follow up assessment.

Treatment Protocol Group I: an oral preparation (capsule) of HA 100 mg, CS 400 mg, N-Acetylglucosamine 200 mg and vitamin C 80 mg once a day in the morning plus an oral preparation of cranberry, D-mannose, propolis extract, tumeric and Boswellia twice a day for three months.

Group C: an oral preparation of cranberry, D-mannose, propolis extract, tumeric and Boswellia twice a day for three months.

After three months of treatment (follow up 1) all women were evaluated with medical and sexual history. Participants also completed the FSFI and IPSS questionnaires. At this point the treatment was reversed (crossover scheme) for additional three months.

At 6 months follow up (follow up 2) participants were again investigated with medical and sexual history and the IPSS and FSFI were completed. Figure 2 report the complete study design. Monthly phone calls were performed to check for adherence to treatment.

Statistics: The sample size consisted of 25 participants in each group, calculated by using the two-sample t-test analysis. Baseline clinical and psychometric scores will be compared between I and C groups. Second, potential differences in FSFI values at 3-6 months follow-up assessment will be evaluated between and within groups. Potential predictors of FSFI improvement will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

sexually active (with at least four occasions of sexual intercourse per month), reproductive-aged (older than 18 years) women with symptomatic rUTIs. Recurrent UTI was defined as more than two symptomatic episodes of uncomplicated UTI within 6 months, or more than three within 12 months

Exclusion Criteria:

* younger than 18, if they had used combined hormonal contraception during the previous 6 months; pregnant, breastfeeding or trying to conceive, if they had symptoms of upper UTI, a history of urinary tract anomalies/vesicoureteral reflux, stress urinary incontinence, interstitial cystitis, diabetes, urinary tract stones, neurologic conditions, clinical depression or depressive symptoms

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Improvement in sexual symptoms | 12 months
  Improvement in sexual symptoms scored with the FSFI questionnaire

SECONDARY OUTCOMES:
Improvement in urinary symptoms | 12 months
  Improvement in urinary symptoms scored with the IPSS questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Ca' Granda Ospedale Maggiore Policlinico, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided
available upon request

REFERENCES:
- [Derived] Boeri L, De Lorenzis E, Lucignani G, Turetti M, Silvani C, Zanetti SP, Longo F, Albo G, Salonia A, Montanari E. Oral preparation of hyaluronic acid, chondroitin sulfate, N-acetylglucosamine, and vitamin C improves sexual and urinary symptoms in participants with recurrent urinary tract infections: a randomized crossover trial. J Sex Med. 2024 Jun 27;21(7):627-634. doi: 10.1093/jsxmed/qdae052. PMID 38721680